CLINICAL TRIAL: NCT06781645
Title: Evaluation of the Effects of Serious Cognitive Games on a Digital Tactile Table for Elderly People with Alzheimer's Disease or Related Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RIVAGES (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2024-A02676-41
Record Dates: First submitted 2024-12-09; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease or Associated Disorder
Keywords: serious games; interactive digital table; Alzheimer disease; Old people; cognitive stimulation
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a randomised crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- programme A, with digital table (Experimental)
  Interventions: Other: The system involves a digital table with a tactile and interactive surface, providing several play areas. It simulates a village and offers different types of serious cognitive games: semantic memory
- programme B, without digital table (No Intervention)

INTERVENTIONS:
Other: The system involves a digital table with a tactile and interactive surface, providing several play areas. It simulates a village and offers different types of serious cognitive games: semantic memory — Each patient included will benefit from a series of 6 sessions of cognitive stimulation with the interactive digital table of cognitive games 'Le Village de Verdurable'©, and a series of 6 sessions of 'classic' weekly cognitive stimulation at the rate of one session per week, i.e. without the digital table and using the methods of cognitive stimulation normally used in the department. The weekly session used as a comparator in the usual condition will be a session based on concentration and attention with target finding or error finding. The order in which these 2 series of 6 sessions will be carried out will be defined randomly (by drawing lots) before the start of the trial.
  Arms: programme A, with digital table

SUMMARY:
Alzheimer's disease and related disorders are chronic, progressive diseases that have a major impact on the lives of sufferers and their families. They lead to a decline in cognitive function and are associated with a loss of independence and quality of life for sufferers. The loss of autonomy associated with major cognitive disorders can lead to feelings of worthlessness and loss of self-esteem. People may feel sad, depressed and, above all, very anxious. When this anxiety is linked to relationships with others, it can become major social anxiety, which aggravates the negative feelings and contributes to the deleterious progression of the neurodegenerative disease. Feelings of low self-esteem and/or the anxiety that accompanies them cannot be treated solely by long-term psychotropic drugs, as these can worsen the disorders through iatrogenesis. In this context, non-drug approaches can be seen as an essential complement.

Cognition-based therapies, including cognitive stimulation, are based on a neuroeducational approach that can be deployed at different stages of the disease, either individually or in groups. Other patient-centred cognitive stimulation techniques have also been developed. In recent years, research has focused on serious digital games, which seem to combine rehabilitation possibilities in a playful form, making it easier for patients to adhere to them. They can also be used to work on motor skills, spatial reference, reflexes and speed and potentially improve verbal and non-verbal learning. Several recent meta-analyses have shown that brain games are an innovative and potentially effective approach to cognitive training for elderly people with cognitive disorders.

Based on the existing literature, experimenting with a serious digital cognitive game could potentially produce beneficial results by improving parameters such as self-esteem and anxiety in patients with early or moderate Alzheimer's disease or a related illness. As part of their weekly cognitive stimulation programme at the day hospital, they plan to use the interactive digital table 'Le Village' ©, which can be used to offer fun exercises on working memory, semantic memory, explicit memory and sensory memory, with game objectives focusing on reaction, reminiscence and dexterity. The digital table simulates a village, allowing 6 people to play simultaneously and interact. This digital table can be used for individual or group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Person aged ≥ 65 years
* A person with Alzheimer's disease or a related disorder established by a full medical diagnosis according to DSM-5 criteria, at a mild to moderate stage defined by a Mini-Mental State (MMSE) ≥ 15/30
* A person who regularly attends the day hospital at Charles Foix Hospital Persons able to give their consent to take part in the study

Exclusion Criteria:

* Person with severe neurocognitive disorders (MMSE < 15/30)
* Person refusing to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rosenberg Self-Esteem Scale | about 3 months
  40-point scale: the higher the score, the higher the self-esteem, and the lower the score, the lower the self-esteem.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | about 3 months
  This 14-item scale gives two scores for anxiety and depression, each out of 21 points. A score of more than 11 indicates anxiety or depression.
the Occupational Therapy Engagement Scale | about 3 months
  This 12-item scale can range from 0 to 36 points. The lower the score, the more difficult it is for the person to engage in therapeutic activities, and vice versa.
scale for rating the person being helped during an interaction with a caregiver | about 3 months
  A 10-item scale, with scores ranging from 10 to 20. The lower the score, the less engaged in the activity, and vice versa.

OTHER OUTCOMES:
the French version of the System Usability Scale | about 1 month
  scale consisting of 10 questions. The score is calculated as a percentage, and the higher the score, the more positive the user experience.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Botto R, Callai N, Cermelli A, Causarano L, Rainero I. Anxiety and depression in Alzheimer's disease: a systematic review of pathogenetic mechanisms and relation to cognitive decline. Neurol Sci. 2022 Jul;43(7):4107-4124. doi: 10.1007/s10072-022-06068-x. Epub 2022 Apr 23. PMID 35461471
- [Background] Zhao QF, Tan L, Wang HF, Jiang T, Tan MS, Tan L, Xu W, Li JQ, Wang J, Lai TJ, Yu JT. The prevalence of neuropsychiatric symptoms in Alzheimer's disease: Systematic review and meta-analysis. J Affect Disord. 2016 Jan 15;190:264-271. doi: 10.1016/j.jad.2015.09.069. Epub 2015 Oct 24. PMID 26540080